CLINICAL TRIAL: NCT07313735
Title: The Effect of Cartoon Character-Printed Band Use During Burn Dressing on Fear, Stress, Pain, and Physiological Parameters in Children: A Randomized Controlled Trial
Acronym: CALM-BURN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Rıdvan Akdogan, Assist. Prof. (PhD), Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YUZUNCU_YIL_UNIVERSITY_cartoon
Record Dates: First submitted 2025-12-10; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Burns; Pain, Procedural; Stress, Psychological; Fear; Child; Bandages
Keywords: Burn dressing; Distraction techniques; Cartoon character bandages; Nonpharmacological pain management; Pediatric nursing
MeSH Terms: conditions — Burns; Pain, Procedural; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, parallel assignment design. Eligible pediatric burn patients are randomly allocated into two groups using the Urn randomization method to ensure balanced distribution. This method will involve two parameters (α and β) represented by two different colored balls. The white ball will represent the intervention group, and the blue ball will represent the control group. The intervention group will receive burn dressing using cartoon character-printed adhesive bands, while the control group will receive standard plain adhesive bands. Both groups will undergo the same dressing procedures performed by trained nurses. Outcomes related to fear, stress, pain, and physiological parameters will be measured before, during, and after the intervention to evaluate the effects of the cartoon-printed bands.
Masking Description: This is an open-label study. Participants, care providers, and outcome assessors will be aware of group allocation due to the visible appearance of the cartoon character-printed bands used during the burn dressing procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cartoon character-printed band (Experimental): Children receiving burn dressing with cartoon character-printed elastic bands.
  Interventions: Other: Cartoon-printed band application
- Standard Band Group (Active Comparator): Children receiving burn dressing with standard plain elastic bands.
  Interventions: Other: Standard band application

INTERVENTIONS:
Other: Cartoon-printed band application — Colorful cartoon character-printed elastic adhesive bands will be applied during a single burn dressing procedure. The bands will be applied by the researcher nurse immediately before and throughout the burn dressing process and will remain in place for the entire duration of the dressing procedure. This intervention will be applied during one burn dressing session in the study period to reduce fear, pain, stress, and physiological responses in children.
  Arms: Cartoon character-printed band
Other: Standard band application — Children in this group will receive burn dressing using standard plain elastic adhesive bands. The bands will be applied by the researcher nurse immediately before and throughout a single burn dressing procedure and will remain in place for the entire duration of the dressing process. No additional distraction or visual intervention will be provided during the procedure.
  Arms: Standard Band Group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of using cartoon character-printed medical bands during burn dressing procedures on children's fear, stress, pain, and physiological parameters. Burn dressing is often a distressing and painful procedure for pediatric patients, which may lead to increased anxiety, physiological instability, and negative treatment experiences.

In this study, child-friendly cartoon-printed adhesive bands are used as a non-pharmacological intervention to provide distraction and emotional comfort during burn dressing. By incorporating familiar and visually engaging designs, the intervention seeks to reduce children's perception of pain, alleviate stress, and improve physiological stability (heart rate, oxygen saturation, and respiratory rate) during the procedure.

Participants will include children aged 7-11 years receiving burn care in a pediatric burn unit. They will be randomly assigned to either the intervention group (cartoon-printed band use) or the control group (standard plain band use). Fear, pain, and stress will be assessed using validated scales before, during, and after the dressing procedure. Physiological parameters will be measured using a pulse oximeter.

The study is expected to contribute to the development of child-centered, non-pharmacological methods that make medical procedures less stressful and more tolerable for pediatric patients. Results may guide the design of more comforting and engaging treatment environments in pediatric burn care.

DETAILED DESCRIPTION:
Burn injuries are among the most common causes of hospitalization in children and often require repeated painful dressing changes. These procedures can provoke significant fear, stress, and pain, negatively affecting children's cooperation, recovery, and overall treatment experience. Traditional approaches to pain management in burn care frequently rely on pharmacological methods, which may have limitations or adverse effects. Therefore, complementary, non-pharmacological interventions are needed to support children during painful procedures.

The CARE-BURN Trial investigates the impact of using cartoon character-printed adhesive bands as a simple, visual, and child-friendly distraction tool during burn dressing. The intervention is designed to create a more comforting and engaging environment for the child by integrating familiar cartoon images into the medical materials. The visual appeal of the bands is expected to distract children's attention from the painful stimulus, enhance their sense of security, and reduce anxiety and perceived pain intensity.

This randomized controlled study includes children aged 7-11 years who are receiving inpatient or outpatient burn treatment. Participants will be randomly assigned using the Urn randomization method to one of two groups:

Intervention Group: Dressing with cartoon character-printed adhesive bands

Control Group: Dressing with standard plain adhesive bands

Measurements:

Children's Fear Scale (CFS)

Wong-Baker FACES Pain Rating Scale

Perceived Stress Scale for Children (PSS-C)

Physiological parameters: heart rate, oxygen saturation, and respiratory rate

Assessments will be conducted at three time points: before, during, and after the dressing procedure. All data will be collected by trained researchers using standardized procedures.

The expected outcomes include decreased levels of fear, stress, and pain, as well as improved physiological stability among children in the intervention group compared to the control group.

The CARE-BURN study aims to demonstrate that low-cost, visually appealing, and child-centered materials can enhance the comfort and cooperation of pediatric patients during invasive or painful treatments. This approach may provide practical insights for pediatric nurses and healthcare providers seeking to humanize burn care and reduce children's distress during routine medical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 11 years at the time of enrollment.
* Hospitalized children diagnosed with superficial partial-thickness or deep partial-thickness burns (second-degree burns).
* Total Burned Body Surface Area (TBSA) ≤ 10%, calculated using the Rule of Nines or Lund-Browder chart.
* Burn location limited to upper extremities, lower extremities, or trunk.
* Scheduled to undergo routine burn dressing procedures in the pediatric ward.
* Ability of the child to communicate pain and anxiety verbally.
* Written informed consent obtained from parent or legal guardian, and assent from the child when appropriate.

Exclusion Criteria:

* Children with full-thickness (third-degree) or fourth-degree burns.
* Burns involving the face, scalp, neck, or genital region.
* TBSA > 10%.
* Presence of cognitive impairment, developmental delay, or neurological disorder that may interfere with outcome assessment.
* Presence of chronic pain conditions or regular use of analgesics unrelated to burn treatment.
* Initial burn dressing performed in an intensive care unit (ICU).
* Refusal of the child or parent/legal guardian to participate.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Fear Level Assessed by the Children's Fear Scale | Baseline (immediately before burn dressing) and immediately after burn dressing procedure
  Assessed using the Children's Fear Scale . Measures the level of fear experienced by children during burn dressing procedures, scored from 0 (no fear) to 4 (highest fear).

SECONDARY OUTCOMES:
Stress Level Assessed by the Perceived Stress Scale for Children (PeSSKi) | Baseline (immediately before burn dressing) and immediately after burn dressing procedure
  Assessed using the Perceived Stress Scale for Children (PeSSKi, ages 7-11). Measures children's perceived stress during the procedure, scored on a 5-point Likert scale, with higher scores indicating higher stress.
Pain Intensity Assessed by the Wong-Baker Faces Pain Scale | Baseline (immediately before burn dressing) and immediately after burn dressing procedure
  Assessed using the Wong-Baker Faces Pain Scale. Measures self-reported pain intensity, scored from 0 (no pain) to 10 (worst pain).
Heart Rate During Burn Dressing | Baseline (immediately before burn dressing) and during burn dressing procedure
  Heart rate measured using a bedside monitor as an indicator of physiological stress response.
Respiratory Rate During Burn Dressing | Baseline (immediately before burn dressing) and during burn dressing procedure
  Respiratory rate measured as breaths per minute to assess physiological stress.
Oxygen Saturation During Burn Dressing | Baseline (immediately before burn dressing) and immediately after burn dressing procedure
  Peripheral oxygen saturation measured using pulse oximetry to assess physiological response.
Body Temperature During Burn Dressing | Baseline (immediately before burn dressing) and immediately after burn dressing procedure
  Body temperature measured to evaluate physiological stress response during the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Regional Training and Research Hospital, Van, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from this study, including fear, stress, pain scores, and physiological parameters, will be made available to other researchers upon reasonable request. Data will be accessible for research purposes only, following approval by the principal investigator, and will be shared through secure data transfer methods. A data dictionary and study protocol will also be provided to facilitate secondary analyses.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data (IPD) and supporting documents, including study protocol and data dictionary, will be available from June 2026 (after completion of data collection and initial analyses) and will remain accessible for 5 years.
Access Criteria: Access to the IPD and supporting information will be granted to researchers with a legitimate research proposal approved by the principal investigator. Researchers will be able to access de-identified fear, stress, pain scores, physiological parameters, and associated study documentation through secure data transfer methods. Data will be used solely for scientific research purposes, and a signed data use agreement will be required.